CLINICAL TRIAL: NCT01646684
Title: Phase 1 Study to Evaluate Safety, and Preliminary Efficacy of Pasireotide LAR in Castration Resistant Prostate Cancer
Brief Title: Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Pasireotide LAR in Patients With Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230XDE04; 2010-024399-25 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2019-10

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: Prostate cancer, pasireotide LAR, castration resistant prostatate cancer, CRPC, SOM230 LAR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOM230 (Experimental)
  Interventions: Drug: SOM230

INTERVENTIONS:
Drug: SOM230

SUMMARY:
After failure of initial ADT, addition of an anti-androgen is established to treat castration resistant prostate cancer (CRPC). Substitution of the first anti-androgen and anti-androgen withdrawal results in treatment responses in 25-40% of patients for 4-6 months. A more effective second line treatment after failure of first ADT could prolong the time until the state of symptomatic HRPC, which is currently treated with docetaxel and accompanied by significant side effects. Since the importance of the IGF-signaling in PC is not only indicated by preclinical results but also by clinical efficacy of somatostatin analogs, further clinical research with the new somatostatin analog pasireotide is warranted.

This study is designed to define the maximum tolerated dose (MTD) of pasireotide LAR in patients with castration resistant prostate cancer (CRPC). It also aims for a preliminary efficacy evaluation of pasireotide within the dose expansion part at the MTD. Preliminary efficacy will be assessed by evaluation of different measures of prostate cancer e.g. changes in PSA, disease control rate (RECIST 1.1), symptoms and changes of biomarkers linked to the mode of action of pasireotide LAR. The study will also explore characteristics of patients who might benefit most from this treatment approach

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0 - 2
2. Histologically proven adenocarcinoma of the prostate.
3. Patients with CRPC (castration resistant prostate cancer): advanced or metastatic adenocarcinoma of the prostate.
4. Prior treatment with a GnRH-agonist or GnRH-antagonist for at least 6 months. The medication must not have been changed for at least 3 months prior to start of study treatment.
5. Prior treatment with an anti-androgen (e.g. bicalutamide, flutamide, cyproteronacetate) is allowed but not necessary. Patients treated with anti-androgen must have discontinued anti-androgen for at least 6 weeks prior to start of study treatment.

   1. Dose escalation part only: prior treatment with an anti-androgen and GnRH agonist or antagonist is allowed.
   2. Dose expansion part only: prior concomitant treatment with an anti-androgen and GnRH agonist or GnRH antagonist for ≤6 weeks is allowed (in order to control flare up).
6. Serum testosterone within castration level (<50 ng/dl or < 1,7 nM)
7. Disease progression demonstrated by a rising PSA with or without metastases. PSA ≥2 ng/mL at study entry. Rising PSA is defined as two consecutive rises over a nadir value; the individual measurements are obtained at least 1 week apart.

Exclusion criteria:

1. Dose expansion part only: Secondary hormonal manipulation of prostate cancer (other than GnRH agonist or antagonist) for more than 6 weeks, including concomitant anti-androgens.
2. Prior cytotoxic therapy e.g. with docetaxel, mitoxantrone.
3. Patients who have received radiotherapy of target lesions. Patients who have received local radiotherapy of non-target lesions for local symptom control within the last 4 weeks must have recovered from any adverse effects of radiotherapy before recording baseline symptoms. Lesions treated with locoregional therapies within the last 3 months before study inclusion do not qualify as target lesions.

Additional protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Escalation phase: Frequency of dose-limiting toxicities (DLTs) at each dose level associated with monthly administration of pasireotide LAR during the first two treatment cycles by CTCAE version 4.03. | Day 56
  DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications as defined per study prototol. These will be evaluated according to the CTCAE v4.03.
Expansion phase: Proportion of patients without PSA-progression at 6 months compared to baseline. | 6 months
  Progression is defined as a PSA-increase of at least 25% and an absolute increase of at least 2 ng/ml from a nadir value, confirmed by a second value four weeks later.

SECONDARY OUTCOMES:
Incidence of adverse drug events, overall and by severity and incidence of serious adverse events and laboratory abnormalities | 3 - 6 months
  Adverse events will be coded using MedDRA.
Changes in laboratory assessments, and assessment of physical examinations such as vital signs and electrocardiograms | 3 - 6 months
  Abnormalities according notable criteria (i.e., newly occurring CTC grade 3 or 4 laboratory toxicities) will be identified.
Percentage and absolute changes from baseline values in PSA and IGF-1 | 3 - 6 months
Area Under Curve (AUC) | pre-dose, day 21 post dose
Proportion of patients without progression at 6 months, defined as PSA-progression (see above) and symptomatic progression of disease and/or progression documented by imaging according to RECIST 1.1 | 6 months
  PSA progression is defined as an increase in PSA of at least 25% compared to baseline and an absolute increase of 2 ng/ml or more from a nadir value. Symptomatic progression is defined at the investigator's discretion. Radiological progression is assessed according to RECIST 1.1
Median progression-free survival (PFS) | 3 - 6 months
  Progression-free survival (PFS) is defined as the time from date of start of treatment to date of event defined as the first documented progression or death due to any cause.
Median overall survival (OS) | 6 - 15 months
  Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause.
Disease Control Rate by RECIST 1.1 after 6 months | 6 months
  Disease control rate (DCR) is the proportion of patients with a best overall response of CR or PR or SD.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Tübingen

REFERENCES:
- See also: Results for CSOM230XDE04 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17564